CLINICAL TRIAL: NCT00617266
Title: Tobacco Control Among Business Process Outsourcing (BPO) Employees
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Gauravi Ashish Mishra, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 351
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Tobacco Use Cessation
Keywords: tobacco, cessation, BPO, RCT, KAP
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 Control Group (Active Comparator): Distribution of pamphlets containing information on the hazards of tobacco
  Interventions: Other: Tobacco cessation intervention
- Arm 2 (Experimental): Active Health Education sessions (harmful effects of tobacco addiction) followed by focus group discussion for all BPO employees
  Interventions: Other: Tobacco cessation intervention
- Arm 3 (Experimental): Active Health Education and Tobacco Cessation Programme for tobacco users using Behavioural Therapy only
  Interventions: Other: tobacco cessation intervention
- Arm 4 (Experimental): Active Health Education and Tobacco Cessation Programme for tobacco users using Behavioural and Pharmaco-therapy
  Interventions: Other: Tobacco cessation intervention

INTERVENTIONS:
Other: tobacco cessation intervention — Active Health Education and Tobacco Cessation Programme for tobacco users using Behavioural Therapy only
  Arms: Arm 3
Other: Tobacco cessation intervention — Active Health Education and Tobacco Cessation Programme for tobacco users using Behavioural and Pharmaco-therapy
  Arms: Arm 4
Other: Tobacco cessation intervention — Distribution of pamphlets containing information on the hazards of tobacco
  Arms: Arm 1 Control Group
Other: Tobacco cessation intervention — Active Health Education sessions (harmful effects of tobacco addiction) followed by focus group discussion for all BPO employees
  Arms: Arm 2

SUMMARY:
The Business Process Outsourcing BPO industry has been rapidly expanding in India over the last 10 years. There is a concern regarding issues of health and safety that are unique to this new and developing industry. The lack of reliable and relevant information on which to base the response to this concern poses a challenge for safeguarding the health of BPO employees. Elevated stress levels, shift duties, high work targets, lofty income may force many towards addictions to keep them going.

Use of tobacco, which is very common addiction in India, is associated with several health hazards. Anecdotal evidence suggests that smoking and other forms of addictions are at its peak in the BPO industries. We are conducting a research on the tobacco habits among Business Process Outsourcing (BPO) employees to understand the prevalence of different forms of tobacco addiction and the reasons for initiation and continuation of the habit. We will also offer different interventions as a measure of tobacco cessation.

DETAILED DESCRIPTION:
This is a four arm randomized controlled trial among Business Process Outsourcing (BPO) employees working in four different BPO units. The trial is undertaken with the objective to explore the prevalence of tobacco use in its various forms along with factors responsible for initiation and continuation of the habit. This trial also aims to study the change in the knowledge, attitudes and practices among BPO employees after intervention with different tobacco cessation strategies.

Four BPO units with work force of approximately 200 employees each, with the management and employees that consent to participate in the study will be selected for the trial. The aim and purpose of the study will be explained and a written informed consent form in English will be offered. The employees who are willing to participate in the trial, will be recruited after signing the informed consent form.

The subjects involved in the research will be expected to answer a few questions about their socio-demographic, occupational, medical, risk factor history and some questions to assess their knowledge, attitude and practice regarding tobacco use. Following this the tobacco users will be offered one of the tobacco cessation interventions to help them quit tobacco.

Regular follow-up visits will be conducted through out the period of the study. The same questionnaire as the pre intervention will be repeated post intervention, ten months later to assess change in their knowledge, attitude and practice regarding tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* The study participants will be apparently healthy males and females above 18 years of age working in the selected BPO units in Mumbai.

Exclusion Criteria:

* There will be no minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-04 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
To assess the post-intervention knowledge, attitudes and practices regarding tobacco addiction and the change as compared with the pre-intervention records by analysing the outcome with respect to different intervention strategies. | 18 months

SECONDARY OUTCOMES:
The prevalence of tobacco and alcohol addiction among the BPO employees. | 10 months
The prevalence of addiction to different forms of tobacco products. | 10 months
Analysis of the factors responsible for initiation and continuation of tobacco habit. | 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India